CLINICAL TRIAL: NCT00068263
Title: A Phase I/II Trial to Evaluate Three Dimensional Conformal Radiation Therapy (3D-CRT) Confined to the Region of the Lumpectomy Cavity for Stage I and II Breast Carcinoma
Brief Title: 3-Dimensional Conformal Radiation Therapy In Treating Women With Stage I or Stage II Breast Cancer Previously Treated With Lumpectomy and Axillary Node Dissection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0319; CDR0000316246
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: 3-dimensional conformal radiation therapy delivers a high dose of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: Phase I/II trial to study the effectiveness of 3-dimensional conformal radiation therapy in treating women who have undergone lumpectomy and axillary node dissection for stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the technical feasibility and reproducibility of three-dimensional conformal radiotherapy confined to the region of the lumpectomy cavity in women with stage I or II breast cancer.
* Determine the cosmetic results in patients treated with this regimen.
* Determine the complication rates in patients treated with this regimen.
* Determine the local control rate in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients undergo three-dimensional conformal radiotherapy twice daily for 5 days beginning within 8 weeks after surgery.

Patients are followed at 6 weeks, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 19-46 patients will be accrued for this study within 6.3 to 15.3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * Stage I or II (T1, N0; T1, N1; T2, N0; or T2, N1)
  * Unifocal disease (single focus that can be encompassed by one lumpectomy)
  * The following histologies are eligible:

    * Invasive ductal
    * Medullary
    * Papillary
    * Colloid (mucinous)
    * Tubular
* No invasive or extensive in situ lobular carcinoma or pure ductal carcinoma in situ (DCIS)
* No nonepithelial breast malignancies such as sarcoma or lymphoma
* Previously treated with lumpectomy of a lesion no greater than 3 cm and axillary dissection of at least 6 lymph nodes or a sentinel node biopsy

  * Six surgical clips in place delineating the margins of the tylectomy cavity
  * Negative, inked histologic margins of lumpectomy (greater than 2 mm) OR re-excision specimen available for confirmation
  * Negative mammography post-lumpectomy or post-excision if malignancy-associated microcalcifications were initially present
  * No prior lumpectomy so extensive that the cosmetic result is low or poor prior to radiotherapy
* No more than 3 positive axillary nodes
* No proven multicentric carcinoma (tumors in different quadrants of the breast or tumor separated by at least 4 cm) with other clinically or radiographically suspicious areas in the ipsilateral breast unless negative by biopsy
* No palpable or radiographically suspicious contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes unless nodes are histologically negative
* No extensive intraductal carcinoma, indicated by one of the following according to the Harvard definition:

  * More than 25 % of invasive tumor is DCIS and DCIS is in adjacent breast tissue
  * Intraductal carcinoma with microinvasion
* No previously treated contralateral breast cancer or synchronous ipsilateral breast cancer
* No evidence of suspicious microcalcifications
* No Paget's disease of the nipple
* No skin involvement by disease, regardless of tumor size
* No distant metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* At least 2 years

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Technically suitable for breast radiotherapy
* No collagenous diseases (e.g., systemic lupus erythematosus, scleroderma, or dermatomyositis)
* No other medical condition that would limit life expectancy
* No psychiatric or addictive disorders that would preclude giving informed consent
* No other malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 2 weeks since prior chemotherapy
* No concurrent chemotherapy during and for at least 2 weeks after completion of study therapy

Endocrine therapy

* Concurrent anastrozole or tamoxifen allowed

Radiotherapy

* No prior radiotherapy for the current malignancy

Surgery

* See Disease Characteristics

Other

* No prior nonhormonal therapy for the current malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08; Primary Completion 2005-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vicini, MD, FACR, Study Chair — William Beaumont Hospital - Royal Oak Campus
Locations (2):
- United States (2):
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

REFERENCES:
- [Result] Vicini F, Winter K, Wong J, Pass H, Rabinovitch R, Chafe S, Arthur D, Petersen I, White J, McCormick B. Initial efficacy results of RTOG 0319: three-dimensional conformal radiation therapy (3D-CRT) confined to the region of the lumpectomy cavity for stage I/ II breast carcinoma. Int J Radiat Oncol Biol Phys. 2010 Jul 15;77(4):1120-7. doi: 10.1016/j.ijrobp.2009.06.067. Epub 2009 Nov 10. PMID 19910132
- [Result] Vicini F, Winter K, Straube W, Wong J, Pass H, Rabinovitch R, Chafe S, Arthur D, Petersen I, McCormick B. A phase I/II trial to evaluate three-dimensional conformal radiation therapy confined to the region of the lumpectomy cavity for Stage I/II breast carcinoma: initial report of feasibility and reproducibility of Radiation Therapy Oncology Group (RTOG) Study 0319. Int J Radiat Oncol Biol Phys. 2005 Dec 1;63(5):1531-7. doi: 10.1016/j.ijrobp.2005.06.024. Epub 2005 Sep 29. PMID 16198508
- [Result] Vicini F, Winter K, Straube W, et al.: A phase I/II trial to evaluate three dimensional conformal radiation therapy (3D-CRT) confined to the region of the lumpectomy cavity for stage I/ II breast carcinoma: initial report of feasibility and reproducibility of Radiation Therapy Oncology Group (RTOG) study 0319. [Abstract] Breast Cancer Res Treat 88 (Suppl 1): A-4067, 2004.
- [Derived] Chafe S, Moughan J, McCormick B, Wong J, Pass H, Rabinovitch R, Arthur DW, Petersen I, White J, Vicini FA. Late toxicity and patient self-assessment of breast appearance/satisfaction on RTOG 0319: a phase 2 trial of 3-dimensional conformal radiation therapy-accelerated partial breast irradiation following lumpectomy for stages I and II breast cancer. Int J Radiat Oncol Biol Phys. 2013 Aug 1;86(5):854-9. doi: 10.1016/j.ijrobp.2013.04.005. Epub 2013 May 29. PMID 23726000